CLINICAL TRIAL: NCT07282743
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Tolerability of GL0034 Among Type II Diabetes Mellitus Subjects Who Are Obese or Overweight With Weight-related Comorbidities
Brief Title: Efficacy and Safety of GL0034 in Overweight or Obese Adults With Type II Diabetes Mellitus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTRE-24-01
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1 (Experimental): Dose Up-titration Period: Participants receive GL0034 starting at Dose Level 1 with titration up to Dose Level 2 for approximately 20 weeks
  Maintenance Treatment Period: Once participants reach their final designated doses, they will continue to receive the final designated doses by weekly subcutaneous administration until the end of Week 48.
  Interventions: Drug: GL0034 Dose Level 1; Drug: GL0034 Dose Level 2
- Arm 2 (Experimental): Dose Up-titration Period: Participants receive GL0034 starting at Dose Levels 1 to 3 with titration up to Dose Level 2 for approximately 20 weeks
  Maintenance Treatment Period: Once participants reach their final designated doses, they will continue to receive the final designated doses by weekly subcutaneous administration until the end of Week 48.
  Interventions: Drug: GL0034 Dose Level 1; Drug: GL0034 Dose Level 2; Drug: GL0034 Dose Level 3
- Arm 3 (Experimental): Dose Up-titration Period: Participants receive GL0034 starting at Dose Levels 1 to 4 with titration up to Dose Level 2 for approximately 20 weeks
  Maintenance Treatment Period: Once participants reach their final designated doses, they will continue to receive the final designated doses by weekly subcutaneous administration until the end of Week 48.
  Interventions: Drug: GL0034 Dose Level 1; Drug: GL0034 Dose Level 2; Drug: GL0034 Dose Level 3; Drug: GL0034 Dose Level 4
- Arm 4 (Experimental): Dose Up-titration Period: Participants receive GL0034 starting at Dose Levels 1 to 6 with titration up to Dose Level 2 for approximately 20 weeks
  Maintenance Treatment Period: Once participants reach their final designated doses, they will continue to receive the final designated doses by weekly subcutaneous administration until the end of Week 48.
  Interventions: Drug: GL0034 Dose Level 1; Drug: GL0034 Dose Level 2; Drug: GL0034 Dose Level 3; Drug: GL0034 Dose Level 4; Drug: GL0034 Dose Level 5; Drug: GL0034 Dose Level 6
- Placebo (Placebo Comparator): Dose Up-titration Period: Participants receive sham placebo up titration, once weekly for approximately 20 weeks.
  Maintenance Treatment Period: Participants will continue to receive placebo once weekly through subcutaneous administration until the end of Week 48.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GL0034 Dose Level 1 — Dose 1, once a week
  Arms: Arm 1; Arm 2; Arm 3; Arm 4
Drug: GL0034 Dose Level 2 — Dose 2, once a week
  Arms: Arm 1; Arm 2; Arm 3; Arm 4
Drug: GL0034 Dose Level 3 — Dose 3, once a week
  Arms: Arm 2; Arm 3; Arm 4
Drug: GL0034 Dose Level 4 — Dose 4, once a week
  Arms: Arm 3; Arm 4
Drug: GL0034 Dose Level 5 — Dose 5, once a week
  Arms: Arm 4
Drug: GL0034 Dose Level 6 — Dose 6, once a week
  Arms: Arm 4
Other: Placebo — Placebo, once a week
  Arms: Placebo

SUMMARY:
This is a phase II, randomized, double-blind, placebo-controlled study to evaluate the efficacy and tolerability of GL0034 among type II diabetes mellitus subjects who are obese or overweight with weight-related comorbidities. Subjects will be put on either one of the four treatment arms (GL0034, once a week, subcutaneous injection) or placebo arm (once a week, subcutaneous injection) following initial dose-up titration that takes up to approximately 20 weeks. The primary end point is change in HbA1c levels from baseline (Week 0) to Week 36 following treatments in all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to sign a written ICF or e-ICF.
2. Men or women ≥18 years of age at the time of signing ICF or e-ICF.
3. Participant was diagnosed with type II diabetes mellitus at least 180 days prior to the day of screening.
4. Participant has a HbA1c level of 7.0 - 10.5%, both inclusive, at the time of screening.
5. Participant has a stable BMI ≥27 kg/m2 for at least 90 days prior to screening.
6. Participant is able and willing to undergo fasting blood draw (i.e. at least 8 hours after last eating or drinking) as well as 7-point SMBG check for 3 consecutive days prior to designated scheduled visits by using a home glucometer that is provided by the study site.
7. Participant on stable daily doses of metformin for at least 90 days prior to screening.
8. Participant who are on metformin and not the following agents for at least 3 months prior to screening: DPP-4 inhibitors, alpha-glucosidase enzyme inhibitors, sulfonylureas, sodium-glucose transport 2 inhibitors, amylin analogues, thiazolidinediones, any insulin product, herbals, or ayurvedic agents. Participants are encouraged to follow the standard of care in their study regions, including appropriate diet and lifestyle modifications, rather than make abrupt change in the diabetic management prior to screening without consulting their physicians.
9. If participant is a woman of childbearing potential (WOCP)*, she must agree to use a highly effective method of contraception during the study in conjunction with a barrier method of contraception, and continue the same contraception method at least one months after the last dose of study drug. Highly effective methods of contraception include one of the following: intrauterine device, injectable hormonal contraceptive, contraceptive patch or implant, partner's vasectomy, bilateral tubal occlusion, and sexual abstinence.

   *WOCP includes women who are not surgically sterilized [using hysterectomy/bilateral salpingectomy/bilateral oophorectomy] or post-menopausal [defined as 12 consecutive months of amenorrhea without an alternative medical cause].
10. Male participants with female partners of child-bearing potential must use a barrier method of contraception (e.g., condom) if not surgically sterile (i.e., vasectomy) during the study. In addition, male participants agree to use the same method of contraception for an additional 30 days after the last IP dose and refrain from donating sperm during this period. In the event that the female partner of the male participant becomes pregnant during the study period + 30 days after the last IP dose, an ICF will be provided to the female partner in order to monitor the female partner, pregnancy, and the newborn.
11. If participant is a WOCP, she must have a negative serum pregnancy test (SPT) at Screening and a negative urine pregnancy at baseline, with results available before IP administration.
12. Participant is willing and able to comply with the study protocol, visit schedule, and other study-related instructions and procedures.
13. Participant is willing and able to independently record the response on various scales and make entries using the e-Patient reported outcomes (ePRO) device.

Exclusion Criteria:

1. Participants who have a history of type I diabetes mellitus.
2. A self-reported change in >5% of body weight within 90 days before screening irrespective of medical records.
3. History of pancreatitis (acute or chronic) or >3 hypoglycemic episodes (blood glucose level <70 mg/dL or 3.9 mmol/L) within 90 days prior to screening.
4. Diagnosis of chronic kidney disease with estimated glomerular filtration rate <60.
5. Poorly controlled hypertension with systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg.
6. Poorly controlled hypothyroidism defined as thyroid-stimulating hormone >6 mIU/L or <0.4 mIU/L.
7. Diabetes mellitus and/or obesity that is induced by endocrine disorders (e.g. Cushing Syndrome) or medication use (e.g. corticosteroids) as judged by the Investigator.
8. Previous surgical treatment for obesity (liposuction and/or abdominoplasty performed >1 year before screening is allowed). Previous or planned (during the trial period) obesity treatment with surgery or a weight loss device. However, previous interventions that, due to reversal or removal, does not have any influence on the participant's weight, in the opinion of the Investigator, are allowed.
9. History of major depressive disorder within 2 years before randomization.
10. History of other severe psychiatric illnesses (i.e. schizophrenia, bipolar disorder).
11. Any lifetime history of a suicidal attempt.
12. Participants with any medical condition [i.e. gastroparesis, uncontrolled gastroesophageal reflux disease, or diarrhea with or without a diagnosis of a diagnosis of irritable bowel syndrome] that, in the opinion of the Investigator, can confound study efficacy assessments or safety concerns.
13. Participant had a myocardial infarction, unstable angina pectoris, or ischemic stroke within the past 6 months prior to IP administration.
14. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2, sudden cardiac death, unexplained death, long QT syndrome, or death from a primary dysrhythmia potentially associated with QT prolongation in any family member.
15. Surgery scheduled for the trial duration period, except for very minor surgical procedures in the opinion of the Investigator.
16. Participants with active malignancy.

    Note: participants with past history of malignancy may be included if:
    * Participant has history of basal cell or in-situ squamous cell carcinoma of skin that has been adequately treated and resolved, per Investigator's judgement.
    * Participant has history of other malignancy that have been adequately treated with no evidence of recurrence/relapse within the last 5 years, per Investigator's judgement.
17. Presence of diabetic retinopathy [both nonproliferative diabetic retinopathy and proliferative diabetic retinopathy]) or maculopathy in either eye that was verified by a fundoscopic examination within 90 days prior to screening or during the study.
18. Known moderate to severe coronary, carotid, or peripheral vascular disease that has planned or will likely need revascularization during the study.
19. Participants with any other condition, which in the opinion of the Investigator, precludes participation in the study (either poses an unacceptable risk to the participant or interferes with assessment/interpretation of study outcomes).
20. Known hypersensitivity to the study IP or its excipients.
21. History of alcohol or drug abuse in the previous two years (Alcohol abuse in this study is defined as >14 standard drinks per week in men or >7 standard drinks per week in women ± a history of alcohol withdrawal symptoms ± institutionalized/hospitalized due to alcohol use ± binge drinking with >5 standard drinks on a single occasion in men or >4 standard drinks on a single occasion in women).
22. Participants are taking, or will start, medications with narrow therapeutic index such as digoxin, warfarin, etc, or those that will prolong QTc interval.
23. Participants received any medications for the treatment of type II diabetes mellitus other than those stated in the inclusion criteria within 90 days before screening. Short-term insulin treatment for a maximum of 7 days prior to screening is allowed. Prior insulin treatment for gestational diabetes is also allowed.
24. Participants who have used medications in the family of GLP-1 agonists in the past.
25. Treatment with any herbal diet supplements, over-the-counter diet medications as an attempt to lose weight within 90 days before screening.
26. Treatment with orlistat, lorcaserin, zonisamide, topiramate, phentermine, buproprion, or naltrexone that could promote weight loss within 90 days before screening.
27. Participation in any organized or online weight-reduction program (i.e. Weight Watchers) within 90 days before screening.
28. Screening calcitonin ≥50 ng/L (pg/mL).
29. Participants having clinically significant abnormal values on Screening laboratory tests or other evidence of uncontrolled disease involving any system-organ (e.g., cardiovascular, pulmonary, renal, hepatic, neurological, endocrine, gastrointestinal, psychiatric etc.) that, in the opinion of the Investigator, would put the participant at risk by participating in the study.
30. Participants with positive urine drug screen [amphetamine, barbiturate, benzodiazepine, cocaine, opiates] with substances that are not part of participant's routine medical care. Tetrahydrocannabinols is acceptable for as long as its use is legally allowed by participant 's home state or country.
31. Participants have clinically significant ECG abnormality , including QTcF >450 msec for males and >470 msec for females, or at high risk for arrhythmia such as judged by the Investigator conditions listed in Criteria #13 above, brady-arrhythmias, tachy-arrhythmias, ventricular arrhythmias, torsade de pointes, high-degree atrioventricular block, or New York Heart Association Class III and IV congestive heart failure.
32. Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c levels from baseline (Week 0) to Week 36 following treatments in all participants | Week 36

SECONDARY OUTCOMES:
Number of participants with an HbA1c <7.0%, <6.5%, or <5.7% | Week 36 or Week 48
Change in HbA1c levels from baseline (Week 0) to Week 48 following treatments in all participants | Week 48
Change in HbA1c levels over time from baseline (Week 0) to Week 48 following treatments in all participants | Week 48
Percent change (%) in body weight and BMI from baseline (Week 0) to Week 36, Week 48, and over time from baseline to Week 48 following treatments in all participants. | Week 36 and Week 48
Percent of participants who achieved ≥5%, ≥10%, ≥15%, >20%, >25% weight loss from baseline to Week 36 or Week 48 of treatments in all participants. | Week 36 or Week 48

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Family First Medical Research Center, Hialeah Gardens, Florida
  - GTL Medical & Research Group, Miami, Florida
- India (3):
  - Life Care Hospital and Research Centre, Bangalore, Karnataka
  - Jothydevs Diabetes Research Centre, Trivandrum, Kerala
  - Madras Diabetes Research Foundation (MDRF), Chennai, Tamil Nadu